CLINICAL TRIAL: NCT05200559
Title: The Efficacy of T-regulatory Cell Depletion with E7777 Combined with Immune Checkpoint Inhibitor, Pembrolizumab, in Recurrent or Metastatic Solid Tumors: Phase I/II Study
Brief Title: T-regulatory Cell Depletion with E7777 Combined with Pembrolizumab in Recurrent or Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alexander B Olawaiye, MD (Other)
Collaborators: Dr. Reddys Laboratories, SA (Industry)
Responsible Party: Sponsor-Investigator, Alexander B Olawaiye, MD, Assistant Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCC 21-166
Record Dates: First submitted 2022-01-05; First posted 2022-01-20 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-11

CONDITIONS: Epithelial Ovarian Cancer
Keywords: PD1/PD-L1-based immunotherapy; Immune Checkpoint Inhibitors (ICI); High Microsatellite Instability (MSI-H); Mismatch Repair Deficiency (dMMR)
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Turcot syndrome | interventions — pembrolizumab; E7777 fusion protein; denileukin diftitox

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- E7777 + Pembrolizumab (Experimental): Phase l:
  E7777: Dose Level 1, 3 µg/kg; Dose Level 2, 6 µg/kg; Dose Level 3, 9 µg/kg; Dose Level 4, 12 µg/kg Day 1-3 - given up to 8 cycles (dose-limiting toxicities assessed for first two cycles, only)
  Pembrolizumab: 200 mg, IV on Day 1 (21-day cycle)
  Phase ll:
  E7777: administered on Day 1-3 at Phase 2 Recommended Dose (P2RD); Day 1-3 up to 8 cycles
  Pembrolizumab: 200 mg, IV on Day 1 (21-day cycle)
  Interventions: Drug: Pembrolizumab; Drug: E7777

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab is a humanized monoclonal immunoglobulin (Ig) G4 antibody that inhibits lymphocytes PD-1 receptors, blocking the ligands that would deactivate it and prevent an immune response, allowing the immune system to target and destroy cancer cells.
  Other Names: Keytruda®
Drug: E7777 — E7777 or denileukin diftitox is a recombinant cytotoxic fusion protein composed of the amino acid sequences for diphtheria toxin fragments A and B (Met1-Thr387)-His and for human interleukin-2 (Ala1-Thr133), indicated for the treatment of patients with persistent or recurrent cutaneous T-cell lymphoma (CTCL) whose malignant cells express the CD25 component of the IL-2 receptor.
  Other Names: ONTAK®

SUMMARY:
Epithelial ovarian cancer (OC) is the most lethal gynecologic cancer: nearly 22,000 women are diagnosed with OC in the US annually and 63% are expected to die from their disease. The 5-year overall survival rate is unacceptably low at 20-30%, with > 50% of patients experiencing recurrence of their disease. Recurrent, platinum-resistant OC is characterized by a low response to chemotherapy (<10-15%) and poor prognosis, with overall survival estimated to be <12 months. Thus, there is an urgent need to identify novel therapies to improve outcomes for patients with recurrent, platinum resistant OC. The primary focus in this trial is targeting tumor associated immunosuppressive T-regs with E7777 combined with PD-1 inhibitor, pembrolizumab. This trial will enroll patients with solid tumors in the dose escalation portion and specified cohorts in the dose expansion portion. In the Phase I portion, 18-30 patients will be enrolled. In the dose expansion portion, approximately 40 patients (20 in each cohort) will be enrolled. Given the relatively poor prognosis and limited treatment options for these patients, this population is considered appropriate for trials of novel therapeutic candidates.

DETAILED DESCRIPTION:
Immunotherapy with immune checkpoint inhibitors (ICI) has emerged as a promising option in several solid tumors, given its durable response and low toxicities. However, the durable benefit of ICI as monotherapy is limited to certain cancers like melanoma, or cancer with a deficient mismatch repair system. However, in the majority of cancers the response rate is lower. For example, the response rate to anti-programmed cell death protein 1 (PD-1) monotherapy in recurrent platinum-resistant ovarian cancer (PROC) has been underwhelming, with a range of 8-15%.

E7777 or denileukin diftitox is a recombinant cytotoxic fusion protein composed of the amino acid sequences for diphtheria toxin fragments A and B (Met1-Thr387)-His and for human interleukin-2 (Ala1-Thr133). Denileukin diftitox has been marketed in the US as ONTAK® (Eisai code name E7272) since 1999 and is indicated for the treatment of patients with persistent or recurrent cutaneous T-cell lymphoma (CTCL) whose malignant cells express the CD25 component of the IL-2 receptor.

This open label study will investigate the safety and efficacy of a combined regimen of pembrolizumab with T-regulatory cell depletion and E7777 in patients diagnosed with recurrent or metastatic solid tumors in the second line setting. This study will have 2 stages: dose escalation and dose expansion. In the dose escalation, any solid tumor where pembrolizumab is approved for or felt as an appropriate therapy by treating physician based on prior trials with encouraging activities including (but not limited to): renal cell carcinoma, melanoma, ovarian cancer, MSI-H cancer, endometrial cancer (EC), and non-small cell lung cancer, hepatocellular carcinoma, cervical cancer, urothelial cancer. The expansion cohort will include ovarian cancer and MSI-H cancer cohort. More cohorts can be considered later.

The TITE-CRM method of dose assignment will be used, which will improve the quality of the assessment of potential toxicities better than the 3+3 method, and will facilitate the evaluation of efficacy. Participants will be treated until disease progression or unacceptable toxicities and/or dose limiting toxicities. E7777 will be given for 8 cycles and Pembrolizumab will be continued after that.

ELIGIBILITY:
Inclusion Criteria:

* Ability to comply with the study protocol, in the investigator's judgment
* Histologically or cytologically confirmed solid tumors (cutaneous melanoma, non-small cell lung cancer, renal cell carcinoma, endometrial cancer, ovarian cancer, MSI-H solid tumors (deficient mismatch repair system or other solid tumors) that have progressed on or refractory to standard of care therapies for their disease
* Phase I dose escalation phase

  * Advanced metastatic or recurrent solid tumors (where pembrolizumab is approved and/or have shown efficacy) that have progressed on or refractory to standard of care therapies for their disease
  * Prior anti-PD1 or PDL1 therapy is allowed
  * Prior anti-CTLA4 therapy is allowed if had anti-CTLA4 free interval of 6 months or more
  * At least one prior line of therapy in the dose escalation phase
* Phase Ib dose expansion cohorts

  * Platinum-resistant recurrent ovarian cancer (recurred within 6 months or less of prior platinum therapy) or post-PD1/PDL1 MSI-H cancers (mismatch repair deficient tumors). Patients in the ovarian cancer cohort must have received chemotherapy plus bevacizumab unless bevacizumab is contra-indicated or considered risky per treating physician.
  * Prior 1-5 lines of therapy for dose expansion
  * Prior anti-PD1/PDL1 therapy is allowed in the MSI-H cohort but not in the ovarian cohort
  * Prior anti-CTLA4 therapy is not allowed.
  * Primary platinum- refractory cancers are excluded in the dose expansion (progressed during or within 3 months of primary platinum therapy)
* Measurable disease per RECIST v1.1

  o Previously irradiated lesions can be considered as measurable disease only if progressive disease has been unequivocally documented at that site since radiation.
* Availability of a representative tumor specimen for exploratory biomarker research
* ECOG Performance Status of 0-1
* Life expectancy ≥ 6 months
* Adequate hematologic and end-organ function, defined by the following laboratory test results, obtained within 14 days prior to initiation of study treatment:

  * ANC ≥ 1.5 × 109/L (1500/L) without granulocyte colony-stimulating factor support
  * Platelet count ≥ 100 × 109/L (100,000/L) without transfusion
  * Hemoglobin ≥ 90 g/L (9 g/dL) o Patients may be transfused to meet this criterion.
  * AST, ALT, and alkaline phosphatase (ALP) ≤2.5 × upper limit of normal (ULN), with the following exceptions:

    * Patients with documented liver metastases: AST and ALT ≤ 5 × ULN
    * Patients with documented liver or bone metastases: ALP ≤ 5 × ULN
  * Serum bilirubin ≤1.5 × ULN with the following exception:

    o Patients with known Gilbert disease: serum bilirubin ≤3 × ULN
  * Serum creatinine ≤1.5 × ULN}
  * Serum albumin ≥ 25 g/L (2.5 g/dL)
  * For patients not receiving therapeutic anticoagulation: INR or aPTT × 1.5 × ULN o For patients receiving therapeutic anticoagulation: stable anticoagulant regimen
* Patients with a positive HIV disease are eligible provided they are stable on anti-retroviral therapy, have a CD4 count ≥ 200/μL, and have an undetectable viral load
* No known Hepatitis infection
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods, and agreement to refrain from donating eggs, as defined below:

  * Women must remain abstinent or use contraceptive methods with a failure rate of < 1% per year during the treatment period and for 5 months after the final dose of pembrolizumab and E7777. Women must refrain from donating eggs during this same period.
  * A woman is considered to be of childbearing potential if she is postmenarchal, has not reached a postmenopausal state (≥ 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus). Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices.
  * The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not adequate methods of contraception.
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use a condom, and agreement to refrain from donating sperm, as defined below:

  * With a female partner of childbearing potential or pregnant female partner, men must remain abstinent or use a condom during the treatment period and for 5 months after the final dose of pembrolizumab + E7777 to avoid exposing the embryo. Men must refrain from donating sperm during this same period.
  * The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not adequate methods of preventing drug exposure

Exclusion Criteria:

* Patients who meet any of the following criteria will be excluded from study entry:

  * History of leptomeningeal disease. Patients with brain metastasis are allowed if their brain metastasis was adequately treated with surgery or radiation or both, have been stable for at least 6 months and not on steroids.
  * Uncontrolled tumor-related pain

    * Symptomatic lesions (e.g., bone metastases or metastases causing nerve impingement) amenable to palliative radiotherapy should be treated prior to enrollment. Patients should be recovered from the effects of radiation. There is no required minimum recovery period.
    * Asymptomatic metastatic lesions that would likely cause functional deficits or intractable pain with further growth (e.g., epidural metastasis that is not currently associated with spinal cord compression) should be considered for loco-regional therapy if appropriate prior to enrollment.
  * Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently)

    o Patients with indwelling catheters (e.g., PleurX™) are allowed.
  * Uncontrolled or symptomatic hypercalcemia (ionized calcium > 1.5 mmol/L, calcium > 12 mg/dL or corrected serum calcium > ULN)
  * Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, or multiple sclerosis for a more comprehensive list of autoimmune diseases and immune deficiencies), with the following exceptions:

    * Patients with a history of autoimmune-related hypothyroidism who are on thyroid-replacement hormone are eligible for the study.
    * Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study.
    * Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met:

      * Rash must cover < 10% of body surface area
      * Disease is well controlled at baseline and requires only low-potency topical corticosteroids
      * No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high-potency or oral corticosteroids within the previous 12 months
  * History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan

    o History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
  * Active tuberculosis
  * Significant cardiovascular disease (such as New York Heart Association Class II or greater cardiac disease, myocardial infarction, or cerebrovascular accident) within 3 months prior to initiation of study treatment, unstable arrhythmia, or unstable angina
  * Major surgical procedure, other than for diagnosis, within 4 weeks prior to initiation of study treatment, or anticipation of need for a major surgical procedure during the study
  * History of concurrent second primary malignancy other than the primary cancer within 3 years prior to screening, with the exception of malignancies with a negligible risk of metastasis or death (e.g., 5-year OS rate > 90%), such as adequately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, localized prostate cancer, ductal carcinoma in situ, or Stage I uterine cancer
  * Severe infection within 4 weeks prior to initiation of study treatment, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia
  * Treatment with therapeutic oral or IV antibiotics within 2 weeks prior to initiation of study treatment

    o Patients receiving prophylactic antibiotics (e.g., to prevent a urinary tract infection or chronic obstructive pulmonary disease exacerbation) are eligible for the study.
  * Prior allogeneic stem cell or solid organ transplantation
  * Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the patient at high risk from treatment complications
  * Treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment, or anticipation of need for such a vaccine during pembrolizumab treatment or within 5 months after the final dose of pembrolizumab
  * Has a known history of human immunodeficiency virus (HIV) infection or HIV test (+) in screening test. No HIV testing is required unless mandated by local health authority. Patients with HIV infection with following exception are allowed: HIV-infected patients on effective anti-retroviral therapy with viral load within 6 months of enrollment are eligible for this trial.
  * Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection except following situation: Patients with a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection are allowed to be included if: participant on a stable dose of antiviral therapy, HBV viral load below the limit of quantification. HCV viral load below the limit of quantification.
  * Treatment with investigational therapy within 28 days prior to initiation of study treatment
  * Prior treatment with CD137 agonists or immune checkpoint blockade therapies, including anti-CTLA-4, anti-PD-1, and anti-PD-L1 therapeutic antibodies except what is specified in the inclusion criteria.

    o Prior anti-PD1 or anti-CTLA4 therapy is allowed in the dose escalation cohort and prior PD1/PDL1 inhibitors are allowed in the MSI-H expansion cohort.
  * Treatment with systemic immunostimulatory agents (including, but not limited to, interferon and interleukin 2 [IL-2]) within 4 weeks or 5 half-lives of the drug (whichever is longer) prior to initiation of study treatment
  * Treatment with systemic immunosuppressive medication (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-TNF-α agents) within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during study treatment, with the following exceptions:

    * Patients who received acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy) are eligible for the study after Principal Investigator confirmation has been obtained.
    * Patients who received mineralocorticoids (e.g., fludrocortisone), corticosteroids for chronic obstructive pulmonary disease (COPD) or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal insufficiency are eligible for the study.
  * History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins
  * Known hypersensitivity to Chinese hamster ovary cell products or to any component of the pembrolizumab formulation
  * Known allergy or hypersensitivity to any component of the E7777 formulation
  * Pregnancy or breastfeeding, or intention of becoming pregnant during study treatment or within 6 months for pembrolizumab and E7777 after the final dose of study treatment o Women of childbearing potential must have a negative serum pregnancy test result within 14 days prior to initiation of study treatment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-09-30 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Recommended Phase 2 Dose (RP2D) | Up to 12 months (cohort)
  Dose-limiting toxicities (DLT) related to E7777 with the immune checkpoint inhibitor (ICI), pembrolizumab. DLT per CTCAE v5.0 will be assessed to determine the RP2D of the treatment combination. Up to twenty patients will be evaluated for DLTs during each dose levels for first 2 cycles (42 days). The transition to next dose level will be determined and planned based on the review of the data on the prior dose level. Safety will be assessed by DLTs, as well as the frequency and severity of immune and non-immune mediated adverse events. or a treatment-related toxicity of any grade requiring dose delay of 3 weeks or more between the first and second cycles
Change in T-regulatory cells in tumor | Up to 5 years
  Change in levels of T-regulatory cells within the immune microenvironment of tumors.
Change in CD8+ T cells in tumor | Up to 5 years
  Change in levels of CD8+ T cells within the immune microenvironment of tumors.
Change in myeloid cells in tumor | Up to 5 years
  Change in levels of myeloid cells within the immune microenvironment of tumors.
Change in T-regulatory cells - peripheral blood | Up to 5 years
  Change in T-regulatory cells within the immune microenvironment of peripheral blood.
Change in CD8+ T cells - peripheral blood | Up to 5 years
  Change in levels of CD8+ T cells within the immune microenvironment of peripheral blood.
Change in myeloid cells in peripheral blood | Up to 5 years
  Change in levels of myeloid cells within the immune microenvironment of peripheral blood.

SECONDARY OUTCOMES:
Objective Response | Up to 5 years
  Objective Response will be expressed as the proportion of patients with Complete Response (CR) + Partial Response (PR). Per RECIST v1.1, Complete Response (CR) is defined as disappearance of all target lesions; disappearance of all non-target lesions and normalization of tumor marker level. Partial Response (PR) is defined as at least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD.
Progression-free survival (PFS) | Up to 5 years
  Progression-free survival is the (estimated) median length of time measured from the initial date of treatment to the date of documented progression, or the date of death (in the absence of progression),whichever occurs first, with progression defined by RECIST v 1.1. Progressive disease(PD) is defined as at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions; appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.
Overall survival (OS) | Up to 5 years
  The (estimated) median length of time from the start of treatment that patients remain alive, until death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Olawaiye, MD, Principal Investigator — UPMC Hillman Cancer Center
Locations (1):
- UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mahdi HS, Woodall-Jappe M, Singh P, Czuczman MS. Targeting regulatory T cells by E7777 enhances CD8 T-cell-mediated anti-tumor activity and extends survival benefit of anti-PD-1 in solid tumor models. Front Immunol. 2023 Oct 27;14:1268979. doi: 10.3389/fimmu.2023.1268979. eCollection 2023. PMID 38022532